CLINICAL TRIAL: NCT01858038
Title: Gene Expression During Surgical Scar Remodeling by Fractional Photothermolysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough subjects interested in this study
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, MD, Director of the Wellman Center for Photomedicine, Professor in Dermatology, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010-P-002618
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Hypertrophic Scars
Keywords: Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The scar will be randomized and demarcated as the following: (1) treatment site and (2) control site (no treatment, no intervention) The treatment condition assigned for each site will be kept the same for all following treatment sessions
- Intervention Fractional Laser treatment (Experimental): Intervention: An FDA-approved Fractional 10,600 nm laser source will be used for laser exposures performed 2 months prior to biopsies of treated sites
  Interventions: Device: Fraxel Repair - Fractional Laser treatment

INTERVENTIONS:
Device: Fraxel Repair - Fractional Laser treatment — An FDA-approved Fractional 10,600 nm laser source will be used for laser exposures performed 2 months prior to biopsies of treated sites
  Other Names: Fraxel Repair, Solta Medical, Hayward, CA
  Arms: Intervention Fractional Laser treatment

SUMMARY:
This project aims to understand the molecular biology underlying the improvement of surgical scars treated by ablative fractional photothermolysis (FP). Previous human studies at MGH have shown that FP significantly improves the appearance and functionality of surgical and burn scars. At the Wellman Center, we have conducted a randomized, controlled study on linear surgical scars demonstrating the efficacy of FP to decrease the volume of hypertrophic scars, and to improve the appearance and texture of scars. However, the underlying mechanism of this therapeutic effect is unknown. It is clear that FP induces wound healing and remodeling of the normal skin surrounding microthermal zones (MTZs). Furthermore, other researchers have employed animal models using transgenic zebrafish and the mouse eye, and found that laser treatments induce changes in gene expression in specific cells. We propose to determine whether the effect of FP on scar improvement occurs via changes in patterns of local gene expression within the skin, specifically dermal fibroblasts. By characterizing these changes, we may be able to identify molecular mechanisms that both explain and contribute to the beneficial effects of FP in the surgical and traumatic scar. The molecular insights into the therapeutic effects of fractional laser photothermolysis may provide a basis for future therapeutic strategies to improve scar remodeling.

DETAILED DESCRIPTION:
A prospective, open-label study in 10 healthy adults, ages 18-50, with abdominal scars will be pursued at the Clinical Research Unit at Wellman Center for Photomedicine (MGH). A side-by-side comparison of untreated vs. one topical treatment of ablative fractional photothermolysis in qualifying subjects will be made. Ten subjects will receive treatment on randomly-assigned portions of their scars, in addition to non-treated control sites. The primary measures of efficacy are (a) blinded evaluation of scar improvement from standard digital photographs taken before and after the treatments, (b) changes in scar volume (measured by 3D Image system) and/or scar width, and (c) a quantitative characterization of gene expression measured by mRNA expression levels from treated and untreated scars and control sites. The primary measures of side effects are inflammatory and pigmentary outcomes assessed by blind evaluation of digital photographs taken before and after the treatments. Another study endpoint includes histopathological examination and comparison of treated and untreated scars.

An FDA-approved 10600 nm Fractional laser source will be used for laser exposures performed 2 months prior to 2 skin biopsies (each 24 mm x 4 mm) of treated and untreated scar sites. A control site, with no treatment will also be left for clinical, histological and molecular examination.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are healthy with ages between 18 and 50 years.
2. Subjects who have had their most recent abdominal procedure at least 2 years prior to enrollment in study.
3. Subjects with surgical scars with a length greater than 10 cm or 4 inches.
4. Subjects whose scars are either hypertrophic or atrophic but enlarged.
5. Subjects who are willing to participate in the study.
6. Subjects who are willing to receive laser treatment.
7. Subjects who are willing to receive skin biopsies.
8. Subjects who agree and sign an informed consent relating to study procedures.
9. Subjects who are willing to follow the treatment schedule and post-treatment care requirements.
10. Subjects who had not received any topical treatment for scars in the past month, including corticosteroid injections, topical fluorinated corticosteroids or any other laser treatment.
11. Subjects who are willing to avoid topical or systemic scar treatment, including topical over-the-counter (OTC) corticosteroids, during the study period.

Exclusion Criteria:

1. Subjects with underlying skin or other medical conditions that could have an adverse effect on wound healing.
2. Subjects with evidence of infection on area to be treated or elsewhere on body.
3. Subjects with presence of suntan in the area to be treated.
4. Subjects who have had topical/Injected corticosteroids within 1 month of entering the study.
5. Subjects with known anticoagulation or thromboembolic condition.
6. Subjects who are immunosuppressed.
7. Subjects who are unable to comply with treatment, home care, or follow-up visits.
8. Subjects who are pregnant or breast-feeding.
9. Subjects with known autoimmune disease.
10. Subjects who are enrolled in any other clinical trial using systemic medication; or any other treatment that might interfere with this study.
11. Subjects with known diabetes mellitus

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mRNA (messenger ribonucleic acid) expression | at 8 weeks
  Gene array analysis will be performed with the Affymetrix Expression ConsoleTM software, which contains commonly used probe set summarization algorithms, including the MAS5 Statistical algorithm, Probe Logarithmic Intensity Error Estimation (PLIER), and the Robust Multichip Analysis (RMA).
  Additional statistical analysis will be performed using the SPSS statistical package (version 16.0, SPSS Inc., Chicago, IL). All two-tailed values of P < 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Evaluation of Efficacy | 8 weeks and 10 weeks
  Vancouver Scar Scale (VSS) and Matching Assessment Using Photographs and Scars (MAPS) for scars

OTHER OUTCOMES:
Assessing Subject Side-effects and Satisfaction | 8 weeks and 10 weeks
  In this survey, subjects are given a list of the treatment side effects before treatment (Visit 1, 2) and are asked to rate each question on a scale of 1 to 5. After treatment, they are given this specific survey (but specific to the treatment site) at each subsequent visit as a repeated measure of side effects. Because subjects will be blinded to the treatment assignment (though sites may become obvious), they will be asked the question based on the treatment site name. Treatment site assignments will be kept with study investigators.

CONTACTS AND LOCATIONS:
Overall Officials: R.Rox Anderson, MD, Principal Investigator — Massachusetts General Hospital - Wellman Center for Photomedicine - Harvard Medical School; Fernanda H Sakamoto, MD, PhD, Study Director — Massachusetts General Hospital - Wellman Center for Photomedicine - Harvard Medical School
Locations (1):
- Massachusetts General Hospital - Wellman Center for Photomedicine, Boston, Massachusetts, United States